CLINICAL TRIAL: NCT07232966
Title: The Efficacy and Safety of Perirenal Adipose Tissue Modification Therapy by Focused Power Ultrasound for Resistant Hypertension
Brief Title: Perirenal Adipose Tissue Modification Therapy for Resistant Hypertension
Acronym: PATH-RHT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yan Li (Other)
Responsible Party: Sponsor-Investigator, Yan Li, Professor, Doctor of Medicine, Doctor of Philosophy, Shanghai Institute of Hypertension
Organization: Shanghai Institute of Hypertension (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025148
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Resistant Hypertension
Keywords: perirenal adipose tissue; focused ultrasound
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perirenal adipose tissue modification by focused power ultrasound (Experimental): Perirenal adipose tissue modification (PRATM) by focused power ultrasound at both kidneys will be performed after the randomisation of eligible patients. After 1 month, if 24-h BP was uncontrolled and of at least 145/100 mmHg, alisartan /indapamide 240/1.5mg once daily will be replaced by sacubitril alisartan 232/248mg and indapamide 1.5mg once daily. At the 3-month after the treatment, if BP was uncontrolled, amlodipine will be uptitrated to 5mg twice a day. The duration of the follow-up after randomisation will be 6 months.
  Interventions: Procedure: Perirenal adipose tissue modification by focused power ultrasound
- Sham (Sham Comparator): Sham procedure will be performed at both kidneys after the randomisation of eligible patients. After 1 month, if 24-h BP was uncontrolled and of at least 145/100 mmHg, alisartan /indapamide 240/1.5mg once daily will be replaced by sacubitril alisartan 232/248mg and indapamide 1.5mg once daily. At the 3-month after the treatment, if BP was uncontrolled, amlodipine will be uptitrated to 5mg twice a day. The duration of the follow-up after randomisation will be 6 months.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Perirenal adipose tissue modification by focused power ultrasound — Perirenal adipose tissue modification by focused power ultrasound at both kidneys
  Arms: Perirenal adipose tissue modification by focused power ultrasound
Procedure: Sham — Sham procedure of focused ultrasound at both kidneys
  Arms: Sham

SUMMARY:
The goal of this clinical trial is to investigate if focused power ultrasound (FPU) targeted perirenal adipose tissue modification therapy would be effective and safe in treating resistant hypertension. The primary outcome of the study is the difference in the reduction of 24h mean systolic blood pressure between treatment and sham procedure groups 6 months after treatment. The secondary outcomes include the reduction of clinic blood pressure 1, 3, and 6 months after treatment, the reduction of 24h mean blood pressure 1, 3, and 6 months after treatment, and the drug burden of antihypertensive treatment. The safety evaluation includes the incidence of all-cause death, cardiovascular events (stroke and myocardial infarction), renal failure, and other adverse events.

DETAILED DESCRIPTION:
Hypertension is the most common cardiovascular disease. However, the control rate of hypertension in China is very low. Resistant hypertension is defined as uncontrolled blood pressure despite optimal lifestyle modifications and the use of three appropriately tolerated, maximally dosed antihypertensive drugs (including a diuretic), or controlled blood pressure with four antihypertensive drugs. Resistant hypertension is associated with increased cardiovascular risk and poor prognosis.

Previous studies have shown that bilateral perirenal adipose tissue (PRAT) ablation or denervation leads to a long-term blood pressure reduction in spontaneous hypertensive rats. Focused power ultrasound (FPU) targeted PRAT modification therapy is a novel intervention aiming to physically or chemically modify PRAT using ultrasound energy, remove nerve fibers, and treat hypertension. Preliminary feasibility and safety was proved in a pilot study of 20 patients. However, a larger, randomized trial is needed to prove efficacy and long-term safety of the treatment.

Participants with resistant hypertension will be recruited in 10 centers and then to investigate whether PRAT modification therapy by FPU is effective and safe for patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18-75 years old;
2. 24h ambulatory systolic BP ≥130mmHg and <150mmHg, and 24h ambulatory diastolic BP <100mmHg after at least 4 weeks of combined treatment with 3 antihypertensive drugs (including a diuretic);
3. The ultrasound measured inferior perirenal adipose tissue ≥8 cm3 (with the superior-inferior diameter, left-right diameter, and anterior-posterior diameter all needing to be ≥20 mm);
4. Be willing to participate in the trial, and be able to visit doctors by himself or herself;
5. Sign the informed consent form.

Exclusion Criteria:

1. Secondary hypertension;
2. Occurrence of myocardial infarction, malignant arrhythmia, severe renal failure, or stroke within 6 months;
3. Ambulatory BP monitoring was invalid (<70% valid readings, or <20 daytime readings or <7 nighttime readings);
4. Alanine transaminase (ALT), aspartate transaminase (AST), or total bilirubin (TBL) above twice the normal range; eGFR (CKD-EPI) <45mL/min/1.73m2;
5. Type 1 diabetes mellitus or uncontrolled Type 2 diabetes mellitus (glycated hemoglobin ≥8.5%);
6. Single functionally normal kidney or presence of renal malignant tumor;
7. Bilateral skin diseases at renal region that are not suitable for the therapy;
8. Women in pregnancy, lactating, or planning for pregnancy;
9. Other concomitant diseases that are considered not suitable for participation in the trial;
10. Patients have contraindications to angiotensin receptor-neprilysin inhibitor (ARNIs), thiazide-like diuretic drugs, or calcium channel blocker (CCBs);
11. Non-compliant patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — men or women
Enrollment: 220 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in 24h systolic blood pressure at the 6-month after treatment | 6 months after treatment

SECONDARY OUTCOMES:
Reduction in 24h ambulatory systolic/diastolic blood pressure | 1 month after treatment
Reductions in 24h ambulatory systolic/diastolic blood pressure | 3 months after treatment
Reduction in 24h ambulatory diastolic blood pressure | 6 months after treatment
Reduction in clinic systolic/diastolic blood pressure | 1 month after treatment
Reduction in clinic systolic/diastolic blood pressure | 3 months after treatment
Reduction in clinic systolic/diastolic blood pressure | 6 months after treatment
Drug burden of antihypertensive treatment | 6 months after the treatment
  number of drugs * dosage of drugs

OTHER OUTCOMES:
The incidence rate of all-cause death | 6 months after treatment
The incidence of cardiovascular events | 6 months after treatment
The incidence of renal failure | 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China